CLINICAL TRIAL: NCT02413385
Title: Canadian Diabetes Strategy Research Project - HealtheSteps™: Exercise and Healthy Eating Prescriptions to Reduce the Risk of Diabetes in Rural and Remote Communities: A Pilot Pragmatic Randomized Controlled Trial (Project 3).
Brief Title: Evidence-Based Lifestyle Prescription Program: Pilot Study
Acronym: HeSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Robert Petrella, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HealtheSteps3
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Chronic Disease; Sedentary Lifestyle; Overweight
Keywords: lifestyle intervention; physical activity; exercise; eHealth; technology; coaching; healthy eating
MeSH Terms: conditions — Chronic Disease; Sedentary Behavior; Overweight; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HealtheSteps Program (Experimental): 6 month evidence-based lifestyle Rx program: receive lifestyle Rx's for exercise, physical activity (step counts) and healthy eating and set goals around Rx's (in person sessions at set time points during 6-month period); take part in self-directed healthy living activities to achieve Rx's (Months 0-6); access to a suite of health technology support options for additional support and coaching (Months 0-6).
  Interventions: Behavioral: HealtheSteps Program
- Usual-care wait-list control (No Intervention): No active intervention (usual care).

INTERVENTIONS:
Behavioral: HealtheSteps Program — 6-month evidence-based lifestyle Rx program: At set time points over the 6-month period, participants have in-person visits with a HeS coach at the clinic setting. At each in-person session, the participant receives an individualized Rx for exercise, physical activity (step count) and healthy eating. The HeS Coach and participant then engage in a coaching/goal setting conversation to set detailed plans and goals to achieve their prescriptions. Participants independently choose which activities they will take part in to achieve their lifestyle Rx's and goals. In between in-person sessions, the participants have access to a suite of free-of-charge health technology support tools to: a) track their exercise, physical activity, and healthy eating; and b) receive virtual coaching and support.
  Arms: HealtheSteps Program

SUMMARY:
The HealtheSteps™ (HeS) Program is an evidence-based, community-focused, lifestyle prescription (Rx) program, supported by in-person coaching and innovative health technologies. The program improves the health of Canadians and reduces their risk for chronic disease by tackling three major risk factors that are shared across a number of chronic diseases: physical inactivity, sedentary behaviour and poor diet. Each HeS participant receives an individualized healthy living Rx for exercise, physical activity (step counts) and healthy eating, supported by coaching and technology tools to promote long-term health behaviour change. For this study, the investigators will undertake a 6-month pilot pragmatic randomized controlled trial (RCT), conducted within 5 clinic settings in Southwestern Ontario. The primary aim is to conduct an outcome evaluation to determine the effectiveness of the HeS program in helping at-risk individuals increase physical activity levels, improve eating habits, and improve other health behaviours and health indicators.

DETAILED DESCRIPTION:
The HealtheSteps™ (HeS) program was developed to improve the health of Canadians and reduce their risk for chronic disease (CD) and brings together emerging evidence from the areas of physical activity, nutrition, behaviour change, health technologies, and knowledge transfer, and moves knowledge into practice. HeS is an evidence-based, viable, and scalable healthy lifestyle solution to tackle the epidemic of CD in Canada. HeS goes beyond traditional health promotion messaging to give individuals a specific plan of action to improve their health and provides community settings with hands-on training, and resources from study knowledge brokers (KBs) to facilitate program uptake and sustainability. The investigators suggest that a widely available HeS program has the potential to impact the lives of Canadians at-risk for and living with CD; shift practice patterns within Family Health Teams (FHTs), Community Health Centres (CHCs) and clinics; reduce health care costs associated with CD; and inform policy decisions about health resource allocation and human resource planning. A scaled-up HeS program will offer at-risk Canadians an opportunity to actively participate in an evidence-based, community-focused, affordable (no cost to participant), healthy lifestyle program supported by point-of-care coaching and innovative electronic Health (eHealth) technologies.

This study will use a two-arm, pilot pragmatic randomized controlled trial (RCT) design. It will take place within 5 clinic settings in Southwestern Ontario. Following assessment of eligibility and baseline measurements, participants will be individually randomized (1:1; stratified by clinical setting) to either the intervention group (receiving the HeS program) or to the comparison group (usual care wait-list control). The comparison group will be offered to start the HeS program after a 6 month delay. All participants (both intervention and comparison groups) will receive publicly available healthy eating and physical activity materials at baseline. Measurements will be taken at baseline and 6 months in both groups; additional follow-up measurements will be taken in the intervention group only at 12 months and again at 18 months (from baseline). Groups will be compared at 6-months in order to examine effectiveness of the HeS program; further, follow-up to 12 and 18 months will be used to look at maintenance of any changes in the intervention group only.

ELIGIBILITY:
Inclusion Criteria:

* One or more self-reported or measured risk factors for chronic disease including: a) objectively-measured body-mass index of greater than or equal to 25 kg/m2; b) less than 150 minutes of exercise per week; c) greater than 3 hours of sitting per day; d) less than 8 fruit and vegetable servings per day; e) diagnosis of metabolic syndrome or type 2 diabetes
* Clear Physical Activity Readiness Questionnaire (PAR-Q) (i.e., either by answering "No" to all questions or receiving clearance from a healthcare provider)

Exclusion Criteria:

* Unable to comprehend letter of information and consent documentation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Average steps per day | 6 months (plus 12 and 18 months in the intervention group only)
  Measured over 7-day monitoring period using pedometers (Yamax Digiwalker SW200 model)

SECONDARY OUTCOMES:
Total physical activity (metabolic equivalent (MET)-minutes/week) | 6 months (plus 12 and 18 months in the intervention group only)
  From the International Physical Activity Questionnaire - Short Version
Time spent in sedentary activity (minutes/day) | 6 months (plus 12 and 18 months in the intervention group only)
  From the International Physical Activity Questionnaire - Short Version
Eating habits: Total healthful eating score | 6 months (plus 12 and 18 months in the intervention group only)
  Measured by Starting the conversation questionnaire
Eating habits: Fruit and vegetable consumption | 6 months (plus 12 and 18 months in the intervention group only)
  Measured by the modified Dietary Instrument for Nutrition Education questionnaire
Eating habits: Fatty food score | 6 months (plus 12 and 18 months in the intervention group only)
  Measured by the modified Dietary Instrument for Nutrition Education questionnaire
Eating habits: sugary food consumption | 6 months (plus 12 and 18 months in the intervention group only)
  Measured by the modified Dietary Instrument for Nutrition Education questionnaire
Health-related quality of life: self-rated health | 6 months (plus 12 and 18 months in the intervention group only)
  Visual Analogue Scale score measured using questionnaire known as EQ-5D-3L
Resting systolic blood pressure | 6 months (plus 12 and 18 months in the intervention group only)
  Measured using automated blood pressure monitor
Resting diastolic blood pressure | 6 months (plus 12 and 18 months in the intervention group only)
  Measured using automated blood pressure monitor
Weight loss (absolute and percentage) | 6 months (plus 12 and 18 months in the intervention group only)
  Measured using digital weight scale
Waist circumference | 6 months (plus 12 and 18 months in the intervention group only)
  Measured using tape measure
Body mass index | 6 months (plus 12 and 18 months in the intervention group only)
  Calculated from height (stadiometer) and weight (digital weight scale) measurements

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Petrella, MD, PhD, Principal Investigator — University of Western Ontario, Lawson Health Research Institute
Locations (1):
- SJHC Family Medical Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petrella RJ, Koval JJ, Cunningham DA, Paterson DH. Can primary care doctors prescribe exercise to improve fitness? The Step Test Exercise Prescription (STEP) project. Am J Prev Med. 2003 May;24(4):316-22. doi: 10.1016/s0749-3797(03)00022-9. PMID 12726869
- [Background] Petrella RJ, Lattanzio CN, Demeray A, Varallo V, Blore R. Can adoption of regular exercise later in life prevent metabolic risk for cardiovascular disease? Diabetes Care. 2005 Mar;28(3):694-701. doi: 10.2337/diacare.28.3.694. PMID 15735210
- [Background] Petrella RJ, Lattanzio CN, Overend TJ. Physical activity counseling and prescription among canadian primary care physicians. Arch Intern Med. 2007 Sep 10;167(16):1774-81. doi: 10.1001/archinte.167.16.1774. PMID 17846397
- [Background] Petrella RJ, Lattanzio CN, Shapiro S, Overend T. Improving aerobic fitness in older adults: effects of a physician-based exercise counseling and prescription program. Can Fam Physician. 2010 May;56(5):e191-200. PMID 20463260
- [Background] Petrella RJ, Aizawa K, Shoemaker K, Overend T, Piche L, Marin M, Shapiro S, Atkin S. Efficacy of a family practice-based lifestyle intervention program to increase physical activity and reduce clinical and physiological markers of vascular health in patients with high normal blood pressure and/or high normal blood glucose (SNAC): study protocol for a randomized controlled trial. Trials. 2011 Feb 16;12:45. doi: 10.1186/1745-6215-12-45. PMID 21324150
- [Background] Stuckey M, Fulkerson R, Read E, Russell-Minda E, Munoz C, Kleinstiver P, Petrella R. Remote monitoring technologies for the prevention of metabolic syndrome: the Diabetes and Technology for Increased Activity (DaTA) study. J Diabetes Sci Technol. 2011 Jul 1;5(4):936-44. doi: 10.1177/193229681100500417. PMID 21880237
- [Background] Stuckey M, Russell-Minda E, Read E, Munoz C, Shoemaker K, Kleinstiver P, Petrella R. Diabetes and Technology for Increased Activity (DaTA) study: results of a remote monitoring intervention for prevention of metabolic syndrome. J Diabetes Sci Technol. 2011 Jul 1;5(4):928-35. doi: 10.1177/193229681100500416. PMID 21880236
- [Background] Noble E, Melling J, Shoemaker K, Tikkanen H, Peltonen J, Stuckey M, Petrella RJ. Innovation to reduce cardiovascular complications of diabetes at the intersection of discovery, prevention and knowledge exchange. Can J Diabetes. 2013 Oct;37(5):282-93. doi: 10.1016/j.jcjd.2013.07.061. PMID 24500553
- [Background] Kitson AL, Rycroft-Malone J, Harvey G, McCormack B, Seers K, Titchen A. Evaluating the successful implementation of evidence into practice using the PARiHS framework: theoretical and practical challenges. Implement Sci. 2008 Jan 7;3:1. doi: 10.1186/1748-5908-3-1. PMID 18179688
- [Background] Rycroft-Malone J, Harvey G, Kitson A, McCormack B, Seers K, Titchen A. Getting evidence into practice: ingredients for change. Nurs Stand. 2002 May 29-Jun 4;16(37):38-43. doi: 10.7748/ns2002.05.16.37.38.c3201. PMID 12068568
- [Background] Ward V, House A, Hamer S. Knowledge Brokering: The missing link in the evidence to action chain? Evid Policy. 2009 Aug;5(3):267-279. doi: 10.1332/174426409X463811. PMID 21258626
- [Derived] Gill DP, Blunt W, Boa Sorte Silva NC, Stiller-Moldovan C, Zou GY, Petrella RJ. The HealtheSteps lifestyle prescription program to improve physical activity and modifiable risk factors for chronic disease: a pragmatic randomized controlled trial. BMC Public Health. 2019 Jun 28;19(1):841. doi: 10.1186/s12889-019-7141-2. PMID 31253112
- [Derived] Gill DP, Blunt W, Bartol C, Pulford RW, De Cruz A, Simmavong PK, Gavarkovs A, Newhouse I, Pearson E, Ostenfeldt B, Law B, Karvinen K, Moffit P, Jones G, Watson C, Zou G, Petrella RJ. HealtheSteps Study Protocol: a pragmatic randomized controlled trial promoting active living and healthy lifestyles in at-risk Canadian adults delivered in primary care and community-based clinics. BMC Public Health. 2017 Feb 7;17(1):173. doi: 10.1186/s12889-017-4047-8. PMID 28173782
- See also: Improving the health of Canadians with evidence-based lifestyle prescriptions website — http://www.healthesteps.ca